CLINICAL TRIAL: NCT01934868
Title: A Comparison of the Long Term Outcomes of Prolotherapy Versus Interlaminar Epidural Steroid Injections (ESI) for Lumbar Pain Radiating to the Leg
Brief Title: Prolotherapy Versus Epidural Steroid Injections (ESI) for Lumbar Pain Radiating to the Leg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Reuth Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0309-13-HMO-CTIL
Record Dates: First submitted 2013-08-30; First posted 2013-09-04 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2022-01

CONDITIONS: Sciatica; Spinal Stenosis of Lumbar Region; Degeneration of Lumbar or Lumbosacral Intervertebral Disc
Keywords: low back pain; sciatica; spinal stenosis; epidural injections; prolotherapy; sacroiliac pain or dysfunction.; Ligament laxity
MeSH Terms: conditions — Sciatica; Low Back Pain; Spinal Stenosis; Joint Instability | interventions — Glucose; Solutions

STUDY DESIGN:
Intervention Model Description: This is a study comparing prolotherapy treatments with an active control, which happens to be the gold standard treatment for radicular pain.
Masking Description: No masking is possible at this point in time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolotherapy Injections (Experimental): Each patient will be evaluated clinically and the spinal levels to be injected will be decided upon during each visit. The levels to be injected will largely depend on the pain referral patterns. All prolotherapy injections will be performed under ultrasound guidance.
  A prolotherapy solution of 20% dextrose combined with 1% lidocaine will be injected to facet capsular ligaments and interspinous ligaments of the lumbar spine and the posterior sacroiliac ligaments. Six points will be injected in each treatment session. These sessions will be 4 weeks apart.
  Interventions: Drug: prolotherapy solution of 20% dextrose
- Epidural Steroid Injections (ESI) (Active Comparator): Those patients assigned to the ESI group will receive epidural steroid injections with 80mg methylprednisolone and 10mg buvicaine to the interlaminar space. These will be performed 4 weeks apart and under fluoroscopy. The level that will be injected will depend both on the clinical presentation as well as the size of the interlaminar space seen under fluoroscopy.
  Interventions: Drug: Epidural Steroid Injection

INTERVENTIONS:
Drug: prolotherapy solution of 20% dextrose — After verifying the anatomy of the lumbosacral spine under ultrasound, a 9cm 22 gauge needle will be used to inject the prolotherapy solution to each of the points specified. In order to view the needle under ultrasound, a needle at least as thick as 22G is required. In order for the prolotherapy injections to be safe, bone must be contacted in order to avoid nerve damage. At each point a total of 1cc prolotherapy solution will be injected.
  Other Names: Dextrose 20% solution
  Arms: Prolotherapy Injections
Drug: Epidural Steroid Injection — Prior to the epidural injection a local anaesthetic solution of 1% lidocaine will be injected into the relevant subcutaneous and ligamentous interlaminar space. The injectant solution will be comprised of 80mg methylprednisolone combined with 10mg (2cc) 0.5% bupivicaine. The resulting 4cc will be diluted with another 4cc of normal saline giving a total volume of 8cc. A loss of resistance technique will be used and radiocontrast dye will be injected to verify the placement of the needle prior to injecting the steroid solution.
  Arms: Epidural Steroid Injections (ESI)

SUMMARY:
The hypothesis is that in the treatment of low back pain (LBP) radiating to the leg, the long-term results of prolotherapy are more effective than those of the current conventional treatment: epidural steroid injections (ESI). This research will examine the efficacy of prolotherapy injections versus epidural steroid injections for the treatment of low back pain radiating to the leg. This is a randomized, unblinded study, in which patients seen in the principle investigator's pain clinic will be randomly divided to receive treatments from either the experimental, prolotherapy group, or the active control, ESI group.

DETAILED DESCRIPTION:
The primary goal of the study is to investigate the long-term efficacy of prolotherapy for patients with LBP referring to the leg. The secondary goal is to compare this efficacy with that of epidural steroids. The reason for exploring options other than ESI is that the latter have proved to be disappointing. Comprehensive reviews have been written on interlaminar and transforaminal epidurals which basically show poor long-term results of longer than 3 months. In addition, ESI carries risks of neurological damage, epidural hematoma and infection. However, ESI continues to be the most widely used treatment worldwide. Research also shows that with increasing age, there is an increased incidence of ligament laxity, spondylolisthesis and angulation which may in turn lead to nerve impingement and deterioration in function with time. Sprained and strained ligaments are themselves capable of referring pain down the leg even as far as the ankle. Research shows that much of the pain referred down the leg is not from impinged nerve roots but from other soft tissues, such as the above-mentioned ligaments; these must be addressed and treated not only to treat pain but in order to improve function.

The term prolotherapy is otherwise known as proliferative regeneration therapy and is aimed at doing just the opposite of cortisone, namely, to strengthen the structures injected, usually ligaments. Prolotherapy solutions are also used to treat partially torn tendons, as in the case of partial rotator cuff tears. Research on prolotherapy has shown that this treatment mode produces varying results in the treatment of low back pain and carries fewer risks than epidurals. One can infer from this that it may provide a safer and better long-term treatment method than ESI. Yelland's review shows that prolotherapy works for the treatment of LBP if this treatment method is combined with other measures such as exercises or manipulations. In this study, patients with low back pain radiating to the leg will be randomized to receive either epidural steroid injections or prolotherapy injections using a solution made up of 20% dextrose. In light of the results of the research quoted, it was decided to give exercise instructions tailored to every patient's condition. Both patients from the experimental and the control groups will receive this instruction in order to avoid the presence of another confounding variable.

A precondition to being included in the trial is having either a CT or MRI of the lumbar spine within the previous 18 months and not having any of the exclusion criteria cited below. Once included in the trial, patients will be randomized into the study and control groups. All epidural injections will be performed under fluoroscopy, and radiocontrast dye will be injected to verify that the injectate will be given in the correct place. Patients in this group will receive 3 interlaminar epidural steroid injections approximately 4 weeks apart. The solution injected will be made up of 80mg methylprednisolone acetate with bupivacaine. The level injected will depend on the clinical picture.

All of the prolotherapy dextrose injections will be performed under ultrasound guidance. Prolotherapy patients will receive 5 sessions approximately 4 weeks apart. In each session, 6 injections in different areas of the lumbosacral spine and sacroiliac ligaments will be injected with 20% dextrose solution using a 25 gauge spinal needle. The targeted structures include the following: the facet joint capsular ligaments, interspinous ligaments, and some of the sacroiliac ligaments, depending on the clinical assessment. The clinical picture will determine what levels will be injected in each session.

As described below, patients will be assessed prior to the study and after the study regarding their pain and function.

Because several patients fail to improve and continue to suffer from severe pain, it was considered unethical to keep patients in their original grouping and prevent crossover for a period of 12 months.

Crossover will be permitted if all of the following conditions apply:

1. At least 1 month has passed since the last treatment in the original allocation group
2. NRS pain levels are at least 6 out of 10
3. Pain and function have not improved with the originally allocated treatment
4. The patient requests the crossover. Participants will receive the same treatments in the crossover groups as patients who were originally allocated to those groups Therefore, patients who cross over to the epidural side will receive up to 3 epidural injections approximately 1 month apart. Participants who cross over to the prolotherapy grouping will receive up to 5 treatment sessions also approximately 1 month apart.

Follow-up of crossover participants will also be performed in the same manner and by the same independent investigator as for non-cross-over participants at 1, 3, 6 and 12 months after the last crossover treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pain radiating down one or both legs or to the groin of at least 12 weeks' duration
* Patients with disc lesions with radiating pain to the leg(s)
* Mild spinal stenosis

Exclusion Criteria:

* History of back surgery
* Recent history (less than 2 years) of active malignancy
* Recent fracture in the lumbar spine or pelvis of less than 12 months
* Active locus of infection in the body
* Coagulation disorders, and current anticoagulation therapy, excluding aspirin
* Chronic medication with corticosteroids and NSAIDS (which are said to possibly neutralise the effect of prolotherapy) - the latter must be stopped 24 hours prior to the first treatment session
* Recent injection of cortisone for back pain or any other pathology elsewhere in the body- patients must wait 2 weeks before commencement of the study
* Concurrent significant depressive illness or evidence of catastrophisation, fibromyalgia
* Concurrent history of active autoimmune disease or inflammatory joint disease evidence of a peripheral neuropathy

NOTE:

If any of the above illnesses appear during the time of the treatment in any patient, the patient will be withdrawn from the trial as treatment may be detrimental to his or her health. In addition, follow-up is not relevant to compare a diseased patient with any of the above with patients who are free of the above illnesses.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale | 17 months
  Prior to the first treatment session, patients from both groups will fill out a questionnaire (described later) which will begin with an added item at the beginning: the NRS (numerical rating scale) score. This is to ascertain the intensity of pain he or she suffers in the lower back and or leg. This is a score given between 0 and 10 to estimate the subjective level of pain felt. 10 is a score given to the worst possible imaginable pain, and 0 is no pain at all. At 4 points in time: 1, 3, 6 and 12 months after the last treatment session, patients will be telephoned by a nurse trained in pain to assess pain level according to NRS score. The nurse will be an independent and unbiased investigator. Because patients often suffer from several sorts of pain, it must be stressed to the patients that what is being measured is the very same pain that the patient came to be treated for initially, and not another area which may have developed pain at some later point in time.

SECONDARY OUTCOMES:
Oswestry Back Disability Questionnaire Score | 17 months
  At the same times as being asked about the NRS score, patients will be interviewed and the Oswestry Back Disability Questionnaire will be filled out by an independent investigator who is a nurse trained in the field of pain. She will give a score at each of the above time allotments. The maximal score is 50, and assesses general function and activity of daily living. The higher the score, the worse is the function. Questions asked relate to pain level, ability to wash oneself, lift things, walk, sit, stand, interact socially, travel, and have sexual relations. Patients with a score above 20 or more out of 50 are considered to have a significant disability.

OTHER OUTCOMES:
Number of patients suffering from adverse effects | 1 week after a particular procedure
  In the event of an adverse effect developing after either of the procedures, this will be reported immediately to the Health Ministry. Number of adverse effects in both groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Osnat Wende, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Pain Unit, Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: When all of the follow-up is completed - hopefully within 12 months

REFERENCES:
- [Background] Benyamin RM, Manchikanti L, Parr AT, Diwan S, Singh V, Falco FJ, Datta S, Abdi S, Hirsch JA. The effectiveness of lumbar interlaminar epidural injections in managing chronic low back and lower extremity pain. Pain Physician. 2012 Jul-Aug;15(4):E363-404. PMID 22828691
- [Background] Manchikanti L, Buenaventura RM, Manchikanti KN, Ruan X, Gupta S, Smith HS, Christo PJ, Ward SP. Effectiveness of therapeutic lumbar transforaminal epidural steroid injections in managing lumbar spinal pain. Pain Physician. 2012 May-Jun;15(3):E199-245. PMID 22622912
- [Background] Iguchi T, Kanemura A, Kasahara K, Kurihara A, Doita M, Yoshiya S. Age distribution of three radiologic factors for lumbar instability: probable aging process of the instability with disc degeneration. Spine (Phila Pa 1976). 2003 Dec 1;28(23):2628-33. doi: 10.1097/01.BRS.0000097162.80495.66. PMID 14652480
- [Background] Bogduk N. On the definitions and physiology of back pain, referred pain, and radicular pain. Pain. 2009 Dec 15;147(1-3):17-9. doi: 10.1016/j.pain.2009.08.020. Epub 2009 Sep 16. No abstract available. PMID 19762151
- [Background] Cohen SP, Chen Y, Neufeld NJ. Sacroiliac joint pain: a comprehensive review of epidemiology, diagnosis and treatment. Expert Rev Neurother. 2013 Jan;13(1):99-116. doi: 10.1586/ern.12.148. PMID 23253394
- [Background] Yelland MJ, Del Mar C, Pirozzo S, Schoene ML. Prolotherapy injections for chronic low back pain: a systematic review. Spine (Phila Pa 1976). 2004 Oct 1;29(19):2126-33. doi: 10.1097/01.brs.0000141188.83178.b3. PMID 15454703
- [Background] Wilkinson HA. Injection therapy for enthesopathies causing axial spine pain and the "failed back syndrome": a single blinded, randomized and cross-over study. Pain Physician. 2005 Apr;8(2):167-73. PMID 16850071